CLINICAL TRIAL: NCT05653609
Title: A Study Evaluating the Sensitivity and Specificity of the Clinical Classifications Generated by the Cureety Digital Telemonitoring Platform: a Database Study to Validate the Cureety TechCare Algorithm
Brief Title: Sensitivity and Specificity of the Clinical Classifications Generated by the Cureety Digital Telemonitoring Tool
Acronym: POSITEA-VA
Status: Completed | Type: Observational
Sponsor: Cureety (Industry)
Responsible Party: Sponsor
Other Study IDs: CTC-2022-11-A
Record Dates: First submitted 2022-12-01; First posted 2022-12-16 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telemonitoring: Patients monitored by the Cureety digital platform
  Interventions: Device: Cureety TechCare

INTERVENTIONS:
Device: Cureety TechCare — Weekly adverse event questionnaires completed by the patients using a digital tool called Cureety

SUMMARY:
Cureety is a digital telemonitoring platform specifically designed to monitor cancer patients through self-reporting of adverse events, accompany patients and their medical teams and complement existing healthcare practices. The platform aims to detect signs and symptoms of health deterioration and disease progression, allowing the medical team to intervene earlier than usual compared to conventional care.

The patients are asked to respond to an electronic patient-reported outcome (ePRO) questionnaire. The digital tool is configured for each patient that generates specific questions that allow grading of adverse events relevant to their specific treatment and disease profile.

At the core of the platform is the medical device "Cureety TechCare", an algorithm that outputs a "clinical classification" based on the adverse events reported by the patients. There are four levels that correspond to the patients' health states, either "critical" ("red"), "to be monitored" ("orange"), "compromised" ("yellow"), or "correct" ("green"). In the case of a red or orange classification, the patients are asked to contact their medical team. In addition, the medical team can monitor the patient classifications from a distance including receiving notifications when patients are classified red and orange.

The present study was designed to retrospectively evaluate the performance of the "Cureety TechCare" medical device in real-life using data collected in the Cureety database.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older.
* Patients that have completed at least one questionnaire in Cureety
* Patients that have not exercised their right to oppose to the use of their data for clinical research.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be randomly selected from all 1530 patients that used the Cureety telemonitoring platform between the 1st of October 2019 and the 30th of September 2022.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Between the 1st of October 2019 and the 30th of September 2022
  Sensitivity of the medical device to correctly identify patients who are flagged for medical attention

SECONDARY OUTCOMES:
Specificity | Between the 1st of October 2019 and the 30th of September 2022
  Specificity of the medical device to correctly identify patients who are not flagged for medical attention.

CONTACTS AND LOCATIONS:
Locations (1):
- Cureety, Dinan, Brittany Region, France

IPD SHARING:
Plan to Share IPD: Undecided